CLINICAL TRIAL: NCT03021603
Title: A Brief Hope Intervention to Increase the Hope Level and to Improve the Physical and Mental Health of Patients Receiving Palliative Care: a Randomized Controlled Trial
Brief Title: Evaluation on the Effects of a Brief Hope Intervention to the Symptoms in the Palliative Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, CHAN Kitty, Lecturer, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS20160205005
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Psychological
Keywords: Hope; psychotherapy; palliative; low-intensity intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This is a 4-week Brief Hope Intervention
  Four sessions in total:
  two face-to-face sessions (1-hour) and two telephone follow up sessions (30 mins) in between.
  Homework : A booklet is prepared for the participants for reviewing their planned goals and recording achieved targets.
  Interventions: Behavioral: Brief Hope Intervention
- Control Group (Experimental): Standard care:
  Clinic follow up and normal hospital care. Logistic call and social communication On completion of the 4-week standard care, the 4-session brief hope intervention will be offered
  Interventions: Behavioral: Brief Hope Intervention

INTERVENTIONS:
Behavioral: Brief Hope Intervention — The present Brief Hope Intervention (BHI) is a four-weeks individual intervention:
  Hope enhancement strategies included sharing and recalling past successes, hope-based goal mapping exercises, examining possible pathways to reach the targeted goals, hope visualization exercise and positive self-talk.
  Purpose: help participants to develop positive thoughts.
  The programme consists of four sessions:
  Two face-to-face sessions (1-hour) and two telephone follow up (30 mins) Homework: A booklet is prepared for the participants for reviewing their planned goals and recording achieved targets.

SUMMARY:
Aims. This paper describes the study protocol of a manualized brief positive intervention (BHI). In addition, it reports the on the modification of a hope intervention based on the theoretical proposition - hope theory, and its feasibility when applying to palliative cancer and non-cancer patients.

Background. Hope was found to account for therapeutic changes in clients with depressive symptoms or chronic pain. Nevertheless, little is known about the integration of such active ingredients to brief and low intensity psycho-therapeutic interventions to patients receiving palliative care were not adequately tested.

Design. The study included two stages: (1) manual development, and (2) a single blinded randomized controlled trial.

Methods. Participants will be randomly assigned in equal number into either the brief hope intervention or the controlled arm on completion of the baseline assessment. Participants of the intervention group will be receiving the four-week intervention, while those allocated to the control arm will be receiving the routine care and social chats. The intervention is a manualized program that consists of four sessions at weekly intervals (two face to face sessions and two telephone follow up in between). The core content is modified from an eight sessions hope therapy. Expert panel feedback and trial on targeted populations were completed. Four participants received the program to determine its acceptability prior to feasibility testing. The process and practical considerations were evaluated to allow refinement of the program and to ensure the quality of intervention.

Outcome measures comprise of changes in state hope score and the depression scores measured respectively by State Hope Scale and Centre for Epidemiological Study Depression Scale. The secondary outcomes are the common signs and symptoms in cancer patients measured by The Condensed Memorial Symptom Assessment Scale. Data collection will be done prior to the intervention (baseline), immediately and one month after the intervention. Additional use of qualitative interview to explore their experiences in the intervention, including satisfaction with the intervention and the treatment fidelity will be conducted.

DETAILED DESCRIPTION:
Introduction According to the Medical Research Council guidance, there are four critical steps to systematically establish a standardize intervention content and mode of delivery through phased approach. Theory and evidence-based practice, feasibility or piloting to test the procedure, estimate recruitment/retention, determining sample size, evaluation and implementation are the four keys of the best practice described in the guideline. In this article, we reported three steps in developing an evidence-based intervention, namely brief hope intervention that addresses the management of cancer and palliative care patients: (1) preparation of the present program, (2) description of the protocol of the feasibility test, and (3) an experimental study using wait list control design.

Background Hope intervention is grounded on positive psychology and is mapped onto cognitive-behavioral therapy. It aligns with the 2014-2018 Oncology Nursing Society research priorities, which indicated the need for evaluating the efficacy of integrating protective factors, such as hope, to the care delivery to the patient and family caregivers. In a similar vein, growing evidence has shown the increasing needs of quality palliative care for non-cancer patients, who suffer from complex illnesses and progressing to end-of-life. These patients having unpredictable disease trajectories, significant loss and grief, and anticipated death would lead to depression and hopelessness. As such, the intervention should be extended to non-cancer patients in their last phase of life. The goal of health-promoting palliative care is to create a supportive environment and strengthen actions that intervene along the journey of care giving, loss and death and dying. In a systematic review, hope was found to account for therapeutic changes in clients with depressive symptoms or chronic pain. Nevertheless, such active ingredients of the psychotherapy are not standard elements of multi-modal care management. This warrants the field testing of the present brief hope intervention in patients receiving palliative care.

Hope Theory Hope theory is adopted as the framework in the present study, where hope was believed as the central agent to facilitate the change process. It focuses on three core features: (1) goal setting (goals), (2) problem solving (pathways) and (3) positive self-talk (agency). These elements underlie the key hope strategies used in the intervention. By increasing hope level, the likelihood of therapeutic change will be increased. Its current emphasis complemented the traditional cognitive behavioral therapy by shifting the primary focus on positive potentials as the starting point, thereby promoting meaning in life, fostering personal strengths, positive changes and improving well-being.

Some believed that being overly optimistic is harmful. However, nurturing hope was found to be one of the significant elements in staying positive in the coping experiences of Chinese couples living with cancer. Evidence has shown that high-hope individuals were found to be more creative and effective problem solvers. More important, a number of studies have reported the positive effect of hope in newly diagnosed cancer patient, for example, health, quality of life, self-esteem, reduced major cancer symptoms, such as pain, fatigue, cough, and depression in lung cancer patients or promoting positive changes in breast cancer patients. However, many of these researches are cross-sectional surveys or qualitative studies; others are mindfulness-based or spiritual-based interventions where hope is only one of the active components in the program. Whether improving the hopeful state of cancer patients and palliative care patients would lead to better clinical outcomes remains under explored.

Brief Hope Intervention The present study aimed to examine the effectiveness of a brief hope intervention in improving the hope level and the physical and mental health of cancer and non-cancer Hong Kong Chinese patients who are receiving palliative care. This low intensity psychological intervention can be delivered by caregiver such as nurses to address the needs of these patients and to build their mental and/or physical abilities. Additionally, the skills could be streamlined in daily nursing practice and an ongoing self-help strategy. Would brief hope intervention be as effective as the standard session in clinical population?

Optimal Length of Hope Intervention Preliminary evidence was found. Literature showed that the role and value of hope at the early counseling sessions enhanced a literal shift to experience a sense of worthiness. Focused hope intervention (90 minutes) has led to higher level of hope and increase in perceived life meaning. The statistical robustness is supported by the comparable effect sizes achieved by both the eight 2-hours sessions and the 90-minute single session in previous studies on hope therapy. The effect sizes on the agency and pathway hope scale scores were 0.65 and 0.38 respectively in the long intervention, and were 0.43 and 0.38 in the brief interventions. One large scale brief positive psychology intervention with hope-based intervention (single session plus one booster session) recruited 1,734 participants from the community, showed positive significant changes in well-being and family happiness (ES 0.11-0.14) (Zhou et al., 2015). Encouraging results were also demonstrated is other studies, which has tested a brief meaning in life intervention for advanced cancer Chinese patients (2-sessions: 30-60 and 15-30 minutes respectively). It showed improvement in quality of life and existential distress. Wong, Wong, & Chang (2015) also found a four-sessions program (one visit plus three telephone follow up) effective in reducing hospital readmission in community dwelling patients with chronic illnesses. Nevertheless, there is insufficient evidence on the optimal length of hope intervention for cancer and palliative patients that would produce the desired effect. Thus the present study results could underpin effective palliative care provision across a range of services from hospitalization to discharge facilitation.

Aims The primary research question is whether brief hope intervention would improve the hopeful state and reduce physical symptoms and/or depression level of patients receiving palliative care. Fidelity was assured at the design level and in intervention delivery to establish a standardized procedure, skill adequacy and translating the intervention from research into clinical practice.

Intervention Description of the intervention The present Brief Hope Intervention is a four-weeks individual intervention, helping participants to develop positive thoughts through skills in goal setting, problem solving and positive self-talk. The program consists of four sessions in total: two face-to-face sessions (1-hour) and two telephone follow up sessions (30 minutes) in between. This serves to create the momentum and continuity of intervention. The first session is the core intervention and the final face-to-face session is a summary talk. Two telephone follow up will review their progress and encourage the practice of hope exercises. Hope enhancement strategies included sharing and recalling past successes, hope-based goal mapping exercises, examining possible pathways to reach the targeted goals, hope visualization exercise and positive self-talk. A booklet will be prepared for the participants for reviewing their planned goals and recording achieved targets. Successful experiences and solutions to perceived barriers are entered. Such take-home exercise helps to extend the participants' practice of hope-based skills into their daily living.

Design and Randomization This study is a randomized controlled trial. On completion of the baseline assessment and the screening procedure, eligible participants will be randomly assigned in equal number into either a brief hope intervention or the control group using sets of computer-generated random numbers. The research assistant conducting the assessments will be blinded to the treatment type. However, participants are inevitably aware of the conditions they have been randomized to. To reduce expectancy effects of the advantages of the program, the control arm is casted as a social intervention. Figure 1 presented the data collection using the Consolidated Standards of Reporting Trials, which will be done before the commencement of the intervention (Time1), immediately post-intervention (Time2) and one month after the completion of program (Time 3).

Participants Chinese cancer and non-cancer patients in Hong Kong, who have completed the curative treatment regimen (surgery and/or chemotherapy and/or radiotherapy) or not eligible for the aforementioned treatment, but receiving palliative care will be invited to join the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Clinically diagnosed to have cancer or patients receiving palliative care
3. Willing to participate in face-to-face activities and telephone follow up
4. Alert and oriented, able to sustain for approximately one hour of attention and interaction
5. Communicable in Cantonese, able to read and write Chinese
6. Could be reached by phone

Exclusion Criteria:

Patients having one or above of the below conditions will be excluded from the study.

1. Patients who have planned operation or further chemotherapy and/or radiotherapy within three months
2. Patients who are unable to communicate in Cantonese
3. Patient who has hearing deficit
4. Patient who are disoriented, delirious or cognitively impaired
5. Patients who have been or is receiving counseling or psychotherapy
6. Patients who are clinically depressed diagnosed by medical doctors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
State Hope Scale (SHS) | 4 weeks
  The SHS is a self-report instrument consisting of 6 items (Snyder et al., 1996) used to assess the two ongoing hope indices related to the pathways and agency of hopeful thinking. For instance, 'I can think of many ways to reach my current goals'. It takes approximately 5 minutes to complete. It is rated on an 8-point scale with 1 = definitely false and 8 = definitely true.

SECONDARY OUTCOMES:
The Condensed Memorial Symptom Assessment Scale (CMSAS) | 4 weeks
  The CMSAS a an abbreviated version of the short form MSAS-SF (Chinese version). The instrument measures 14 prevalent symptoms and comprises of two subscales: (1) Physical Symptom (CMSAS PHYS -11 items), (2) Psychological Symptom (CMSAS PSYCH - 3 items), and total score of the CMSAS (CMSAS SUM). Physical symptoms included lack of energy, lack of appetite, pain, dry mouth, weight loss, feeling drowsy, shortness of breath, constipation, difficulty sleeping, difficulty concentrating, and nausea. The psychological symptoms include worrying, feeling sad, and feeling nervous. The items were scored on a 5-point Likert scale from 0 = not at all to 4 = very much.

OTHER OUTCOMES:
Center for Epidemiological Studies Depression Scale (CES-D) | 4 weeks
  CES-D is a 20-item self-report scale measures the frequency of occurrence of depressed mood within one week is in a response format of 4-point Likert scale. The four options are 'rarely or none of the time' (less than 1 days); "some or a little of the time' (1-2 days), "occasionally or a moderate amount of the time" (3-4 days); and "most or all of the time" (5-7 days). Total scores ranging from 0 to 60, with higher ratings denoting higher frequency of depressive symptoms.
Healthcare Resource Utilization | 3 months
  Hospital readmission rate, emergency room utilization and mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Chan Kitty, PhD, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: Yes
Publication of results in May 2018